CLINICAL TRIAL: NCT00689754
Title: The Role of Routine Placement of Nasogastric Tube in Patients With Suspected Upper Gastrointestinal Hemorrhage
Brief Title: Efficacy and Safety Study on Nasogastric (NG) Tube in Patients With Upper Gastrointestinal Bleed
Acronym: NG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Silvio Melo, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 102007-022
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Gastrointestinal Hemorrhage; Liver Cirrhosis
Keywords: gastrointestinal hemorrhage; gastrointestinal intubation; endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NGA (Active Comparator): Patients will receive the standard of care to proceed with nasogastric tube placement, aspiration and lavage up to 1L of normal saline
  Interventions: Procedure: nasogastric tube placement
- NO NGA (No Intervention): Patient presenting with Upper GI hemorrhage going straight to endoscopy.

INTERVENTIONS:
Procedure: nasogastric tube placement — standard nasogastric tube placement, aspiration and lavage up to 1L of normal saline
  Arms: NGA

SUMMARY:
Upper gastrointestinal tract hemorrhage (UGIH) remains a major cause of morbidity and mortality . Nasogastric aspiration (NGA) is routinely performed in patients with UGIH to obtain important clinical data and make therapeutic decisions. But routine use of NGA remains controversial with studies reporting its usefulness and its redundant clinical information. Early esophagogastroduodenoscopy (EGD) is recommended by most gastrointestinal societies to allow for risk stratification and to perform endoscopic treatments. The results of the NGA may assist to differentiate between high-risk versus low-risk lesions. Our hypothesis is that presence of NGA can identify lesions that require endoscopic treatment and provides important clinical information to guide the treating physician. In addition, we hypothesized that the results of the NGA influence the clinical decision of the treating physician regarding the prediction of the need for endoscopic therapy. This observational randomized cross-sectional study will enroll consecutive patients with presumed UGIH and randomized them to NGA and no NGA recording its results. All patients will receive an EGD and its results will also be recorded. Subsequently, we will evaluate if the NGA is important in identifying endoscopically significant lesions. The information gained will help guide clinicians evaluating patient with UGIH.

ELIGIBILITY:
Inclusion Criteria:

* Patients older then 21 years-old presenting with actual or reported: Hematemesis, Melena, or Hematemesis and Melena

Exclusion Criteria:

* Refusal to participate
* Severe comorbid conditions making EGD hazardous for the patient, such as myocardial infarction < 3 months with the exception if the myocardial infarction was caused by the UGIH, hemorrhagic or ischemic stroke < 3 months, decompensated congestive heart failure, severe respiratory failure unless the patient is already intubated
* Survival expected to be less than 72h as judged by treating clinician
* Prisoners
* Patient with severe mental illness precluding the ability to obtain informed consent
* Ongoing anticoagulation which can not be reversed secondary to patient safety
* Strongly suspected gastrointestinal perforation
* Recent endoscopy (less than 30 days)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The number of patients predicted accurately to have a treatable lesion | 24h

SECONDARY OUTCOMES:
Complications of nasogastric aspiration and lavage | 24h
Relationship between time to endoscopy and upper gastrointestinal hemorrhage | 24h
Relationship of nasogastric aspirate and lavage with number of units of packed reb blood cells transfused | 24h
Complication of nasogastric tube placement and aspiration in cirrhotics | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Silvio W Melo, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Result] Luk GD, Bynum TE, Hendrix TR. Gastric aspiration in localization of gastrointestinal hemorrhage. JAMA. 1979 Feb 9;241(6):576-8. PMID 310892
- [Result] Peterson WL. Evaluation and initial management of patients with upper gastrointestinal bleeding. J Clin Gastroenterol. 1981;3(Suppl 2):79-84. PMID 6976367
- [Result] Gilbert DA, Silverstein FE, Tedesco FJ, Buenger NK, Persing J. The national ASGE survey on upper gastrointestinal bleeding. III. Endoscopy in upper gastrointestinal bleeding. Gastrointest Endosc. 1981 May;27(2):94-102. doi: 10.1016/s0016-5107(81)73157-2. No abstract available. PMID 6971777
- [Result] Cuellar RE, Gavaler JS, Alexander JA, Brouillette DE, Chien MC, Yoo YK, Rabinovitz M, Stone BG, Van Thiel DH. Gastrointestinal tract hemorrhage. The value of a nasogastric aspirate. Arch Intern Med. 1990 Jul;150(7):1381-4. doi: 10.1001/archinte.150.7.1381. PMID 2196022
- [Result] Basuk PM, Isenberg JI. Gastric lavage in patients with gastrointestinal hemorrhage. Yea or nay? Arch Intern Med. 1990 Jul;150(7):1379-80. No abstract available. PMID 2369238
- [Result] Cappell MS, Scarpa PJ, Nadler S, Miller SH. Complications of nasoenteral tubes. Intragastric tube knotting and intragastric tube breakage. J Clin Gastroenterol. 1992 Mar;14(2):144-7. doi: 10.1097/00004836-199203000-00015. PMID 1556428
- [Result] Levy H. Nasogastric and nasoenteric feeding tubes. Gastrointest Endosc Clin N Am. 1998 Jul;8(3):529-49. PMID 9654567
- [Result] Barkun A, Bardou M, Marshall JK; Nonvariceal Upper GI Bleeding Consensus Conference Group. Consensus recommendations for managing patients with nonvariceal upper gastrointestinal bleeding. Ann Intern Med. 2003 Nov 18;139(10):843-57. doi: 10.7326/0003-4819-139-10-200311180-00012. PMID 14623622
- [Result] Aljebreen AM, Fallone CA, Barkun AN. Nasogastric aspirate predicts high-risk endoscopic lesions in patients with acute upper-GI bleeding. Gastrointest Endosc. 2004 Feb;59(2):172-8. doi: 10.1016/s0016-5107(03)02543-4. PMID 14745388
- [Result] Lee SD, Kearney DJ. A randomized controlled trial of gastric lavage prior to endoscopy for acute upper gastrointestinal bleeding. J Clin Gastroenterol. 2004 Nov-Dec;38(10):861-5. doi: 10.1097/00004836-200411000-00005. PMID 15492601
- [Result] Cappell MS. Safety and efficacy of nasogastric intubation for gastrointestinal bleeding after myocardial infarction: an analysis of 125 patients at two tertiary cardiac referral hospitals. Dig Dis Sci. 2005 Nov;50(11):2063-70. doi: 10.1007/s10620-005-3008-8. PMID 16240216
- [Derived] Rockey DC, Ahn C, de Melo SW Jr. Randomized pragmatic trial of nasogastric tube placement in patients with upper gastrointestinal tract bleeding. J Investig Med. 2017 Apr;65(4):759-764. doi: 10.1136/jim-2016-000375. Epub 2017 Jan 9. PMID 28069629
- See also: UT Southwestern website — http://www.utsouthwestern.edu